CLINICAL TRIAL: NCT04604782
Title: An Open-label, Single-dose, Safety and Pharmacokinetic Study of Regadenoson in Pediatric Patients
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of Regadenoson in Pediatric Patients
Acronym: Rapiscan PIP
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-262-001
Record Dates: First submitted 2020-10-01; First posted 2020-10-27 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Myocardial Ischemia; Coronary Artery Disease
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease | interventions — regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- adolescents aged 12 to <18 years (Experimental)
  Interventions: Drug: Regadenoson
- children aged 2 to <12 years (Experimental)
  Interventions: Drug: Regadenoson
- infants aged 1 to <24 months and who weigh at least 3 kg (Experimental)
  Interventions: Drug: Regadenoson

INTERVENTIONS:
Drug: Regadenoson — Regadenoson (Rapiscan®): Single i.v. bolus dose in stress rest CMR
  Other Names: Rapiscan

SUMMARY:
This is a multi-centre, open-label, single-dose safety, tolerability and PK-pharmacodynamics (PD) study of the vasodilator regadenoson in 3 paediatric age groups for whom a pharmacologic stress perfusion CMR test is clinically indicated; adolescents aged 12 to <18 years (Cohort A), children aged 2 to <12 years (Cohort B), and infants aged 1 to <24 months and who weigh at least 3 kg (Cohort C). Regadenoson will be used as the pharmacologic stress agent in this study with MPI serving as both surrogate pharmacodynamic marker of the agent (MPR, MBF) and a clinically evaluable examination for the patient

DETAILED DESCRIPTION:
This is a multi-centre, open-label, single-dose safety, tolerability and PK-pharmacodynamics (PD) study of the vasodilator regadenoson in 3 paediatric age groups for whom a pharmacologic stress perfusion CMR test is clinically indicated; adolescents aged 12 to <18 years (Cohort A), children aged 2 to <12 years (Cohort B), and infants aged 1 to <24 months and who weigh at least 3 kg (Cohort C). Regadenoson will be used as the pharmacologic stress agent in this study with MPI serving as both surrogate pharmacodynamic marker of the agent (MPR, MBF) and a clinically evaluable examination for the patient.

At least 54 paediatric patients will be enrolled at approximately 10 centres in Europe: at least 24 adolescents aged 12 to <18 years (Cohort A), at least 18 children aged 2 to <12 years (Cohort B), and at least 12 infants aged 1 to <24 months (Cohort C). The study will be conducted in facilities appropriate for children, and by personnel knowledgeable and skilled in working with paediatric patients. Every attempt will be made to minimise the discomfort of the procedures to the patients. General anaesthesia/sedation with no oral-intake instructions may be used in accordance with age / disease specific requirements of the patient and as deemed necessary by the investigator per standard of care / local practice. In addition, adequate resuscitation equipment and personnel trained and certified in advanced life support must be readily available when regadenoson is administered. A Data Safety Monitoring Board (DSMB) will be in place, and will formally review all safety, efficacy, PK and PD information during the conduct of the study to ensure the safety of patients.

The study will be performed in a sequential manner across the 3 age groups, by decreasing age from adolescents (Cohort A) to children (Cohort B) and to infants (Cohort C). Dosing recommendations for the paediatric population are based on effective dose levels and PK data in adults. Based on a fixed dose of 400 µg regadenoson administered to adults with a mean body weight of 83.8 kg (body weight range: 42 to 161 kg), the effective mean weight-based dose was 4.8 µg/kg (range: 2.5 to 9.5 µg/kg). Within each age group, dosing will be extrapolated from PK-PD data obtained in adults and will be based on body weight-categories to provide approximately the same exposure as 400 µg in adults. The study will start with Cohort A (adolescents). Before the start of dosing in Cohort B, all safety, PK, and PD data obtained in Cohort A will be reviewed by the DSMB. Before the start of dosing in Cohort C, all safety, PK, and PD data obtained in Cohorts A and B will be reviewed by the DSMB.

ELIGIBILITY:
Inclusion Criteria:

* * Male or female adolescent aged from 12 to <18 years (Cohort A) or child aged from 2 to <12 years (Cohort B) or infant aged from 1 to <24 months (Cohort C).

  * Patient weighs at least 3 kg.
  * Patients who need to undergo a clinically indicated pharmacologic stress perfusion CMR test and who are considered fit for a pharmacological stress perfusion CMR by the investigator. The pharmacologic stress perfusion CMR may be performed in patients for further evaluation of cardiovascular conditions or diseases, such as, but not limited to, Kawasaki disease, congenital heart diseases, congenital coronary abnormalities, and post-cardiac surgery / transplantation, etc.
  * Stable medication regimen for at least 7 days prior to dosing. Stable is defined as no addition, discontinuation, or change of any medications (or their doses), that could alter the rate-pressure product (HR x BP).
  * Patients and those whose parents or legally authorised representatives are, in the Investigator's view, likely to be compliant and complete the study will be eligible to participate
  * Post-menarchal female patients must have a negative urine pregnancy test at screening and at pre-dose on the dosing day.
  * Post-menarchal female patients must be practicing abstinence, or be using an effective form of birth control (e.g., intrauterine device, oral contraceptives, contraceptive implants or injections, diaphragm with spermicide, cervical cap, or consort use of condom) for at least 30 days before being enrolled in the study

Exclusion Criteria:

* * Prior allergic reaction to Gd contrast agents and/or regadenoson or any component of its formulation, or to aminophylline or to its components (ethylenediamine and theophylline).

  * Standard clinical contraindications to MRI as per institutional guidance, including patients with cochlear implants and implanted cardiac devices, or considered unfit for a pharmacologic stress perfusion CMR test by the investigator.
  * All patients will be screened for eGFR within 24 hours before the exam and patients presenting with eGFR <30 mL/min/1.73 m2 (by the Schwartz formula) will be excluded.
  * Pregnant or lactating females, or females of childbearing potential not using an acceptable form of birth control (negative urine pregnancy test also required).
  * In the judgment of the Investigator, any clinically significant ongoing medical condition (e.g., myocardial infarction, or unstable angina within 5 days, pericardial inflammatory disease, severe cardiac outflow tract obstruction, acutely decompensated heart failure, uncontrolled epilepsy, high risk for seizures, etc.) or clinically significant laboratory abnormality that is considered to potentially jeopardise the patient's safety.
  * Patients with 2nd or 3rd degree atrioventricular block or sick sinus syndrome with or without an artificial pacemaker.
  * Known or suspected bronchoconstrictive and bronchospastic lung disease either being unstable or requiring active treatment (e.g., wheezing noted on physical exam, frequent exacerbations or active treatment with a bronchodilator or corticosteroids).
  * Out of acceptable range sitting or semi-recumbent resting BP or HR (beats per minute [bpm]) at screening as provided below:

    1. Acceptable range for BP (systolic / diastolic mmHg):
* For Cohorts A and B: 85-130 / 45-90
* For Cohort C: 80-120 / 40-80 b) Acceptable range for HR:
* For Cohort A: 55 to 100 bpm
* For Cohort B: 60 to 120 bpm
* For Cohort C: 70 to 160 bpm

  * Use of any experimental or investigational drug or device within 30 days prior to dosing with study drug
  * Consumption of methylxanthine-containing products such as caffeinated coffee, tea, caffeinated soft drinks, cocoa or chocolate in the 48 hours prior to dosing
  * Aminophylline or theophylline use within 24 hours, dipyridamole use within 48 hours prior to dosing.
  * History of alcohol abuse or drug addiction, as determined by the Investigator
  * Currently smokes more than 5 cigarettes or equivalent per day, and if eligible for the study, would not be able to abstain from smoking from midnight prior to dosing until the end of the study period
  * Positive urine drug screen at the screening visit, including amphetamines, barbiturates, cannabinoids, cocaine, ethanol and opiates. This will be performed for all patients in Cohort A and those patients at age-appropriate risk in Cohorts B and C, as determined by the investigator.

Note: If the patient is currently receiving prescribed medications containing any of these ingredients, re-screening can only be considered if found acceptable based on the best medical judgement of the investigator and after discussion with the medical monitor. Otherwise, patients with a positive urine drug test will be considered a screen failure.

Ages: 4 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Adverse Events (AEs) following administration of Regadenoson | 70 hours after Regadenoson administration
  An overall summary of AEs, SAEs, and Regadenoson-emergent AEs will be presented, coded using the Medical Dictionary for Regulatory Activities (MedDRA) and summarized by system organ class and preferred term.
Changes in physical examinations following administration of Regadenoson | Baseline and 2 hours after Regadenoson administration
  The number of patients with changes in physical examination status from normal at baseline to abnormal at each post-administration time point will be summarized.
Changes in physical examinations following administration of Regadenoson | Baseline and 2 hours after Regadenoson administration
  The percentage of patients with changes in physical examination status from normal at baseline to abnormal at each post-administration time point will be summarized.
Changes in oxygen saturation following administration of Regadenoson | Baseline, 15 and 5 minutes before Regadenoson administration and 1, 3, 6, 10, 15, 30 minutes and 1, 2 hours after Regadenoson administration
  The occurrence of post-administration vital sign values outside the normal limits will be summarized.
Changes in blood pressure in mmHg following administration of Regadenoson | Baseline, 15 and 5 minutes before Regadenoson administration and 1, 3, 6, 10, 15, 30 minutes and 1, 2 hours after Regadenoson administration
  The occurrence of post-administration vital sign values outside the normal limits will be summarized.
Changes in heart rate as bpm following administration of Regadenoson | Baseline, 15 and 5 minutes before Regadenoson administration and 1, 3, 6, 10, 15, 30 minutes and 1, 2 hours after Regadenoson administration
  The occurrence of post-administration vital sign values outside the normal limits will be summarized.
Changes in body temperature (as degree C) following administration of Regadenoson | Baseline and 2 hours after Regadenoson administration
  The occurrence of post-administration body temperature values outside the normal limits will be summarized by counts and percentages by age group and actual dose.
Change from baseline in the results of 12-lead electrocardiograms (ECGs) following administration of Regadenoson | Baseline, 1 and 2 hours after Regadenoson administration
  Descriptive statistics will be used to describe the observed values and change from baseline for ECG intervals (RR, QT, QTcF[Fridericia])
Changes in serum chemistry following administration of regadenoson | Baseline and 2 hours after Regadenoson administration
  The occurrence of post-administration clinical laboratory values outside the normal limits will be summarized.
Time changes of regadenoson blood concentrations (ng/mL) with a single, body-weight adjusted i.v. dose in 3 paediatric populations: adolescents 12 to <18 years,children 2 to <12 years, and infants 1 to <24 months, and who weigh at least 3kg. | 1, 3, 5, 10, and 20 minutes and 1 and 2 hours post Regadenoson administration
  Blood samples for PK assessment will be collected and processed for measurement of Regadenoson blood concentrations. Concentration-time profiles will be evaluated using compartmental methods and a population approach with mixed-effect modelling. A summary will be listed by patient and summarized by age group and actual dose at each time point.

SECONDARY OUTCOMES:
Determine the correlation between regadenoson PK concentration (ng/mL) and changes in HR (bpm), including impact of patient factors. | 1, 3, 5, 10, and 20 minutes and 1 and 2 hours post Regadenoson administration
  The correlation between regadenoson PK concentration and change in HR at different time points will be evaluated using compartment methods and a population approach with mixed-effect modelling adjusted for patient factors.
Determine the associated myocardial hyperaemic response after administration of regadenoson using dynamic first-pass perfusion magnetic resonance imaging (MRI). | 1 hour post Regadenoson administration.
  The Myocardial perfusion reserve (MPR) and Myocardial blood flow (MBF) values derived from the quantitative image analysis of the myocardial perfusion images will be listed per patient and summarized with descriptive statistics by age group and actual dose.
Determine the associated myocardial hyperaemic response after administration of regadenoson using dynamic first-pass quantitative myocardial perfusion reserve (MPR) analysis. | 1 hour post Regadenoson administration.
  The Myocardial perfusion reserve (MPR) and Myocardial blood flow (MBF) values derived from the quantitative image analysis of the myocardial perfusion images will be listed per patient and summarized with descriptive statistics by age group and actual dose.

CONTACTS AND LOCATIONS:
Overall Officials: David Thompson, MD, PhD, Study Director — GE Healthcare
Locations (5):
- Paris Public Hospitals System; Necker Hospital for Sick Children, Paris, France
- Mitera Hospital, Athens, Greece
- Bambino Gesu Children Hospital, Roma, Italy
- United Kingdom (2):
  - Bristol Royal Hospital for Children, Bristol
  - King's College London, Rayne Institute, London